CLINICAL TRIAL: NCT00104637
Title: A Double-blind, Placebo-controlled, Crossover Study of Sildenafil in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Sildenafil for Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kawut, Steven, MD (Individual)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1022
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Results first posted 2012-05-21 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Emphysema
Keywords: Chronic Obstructive Pulmonary Disease; Emphysema; Phosphodiesterase inhibitors; Sildenafil; Exercise testing; Quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil / Placebo (Active Comparator): Sildenafil first, followed by washout, followed by placebo
  Interventions: Drug: sildenafil citrate; Drug: Placebo
- Placebo / Sildenafil (Placebo Comparator): Placebo first, followed by washout, followed by Sildenafil
  Interventions: Drug: sildenafil citrate; Drug: Placebo

INTERVENTIONS:
Drug: sildenafil citrate — sildenafil citrate 25 mg by mouth thrice daily (po tid)
Drug: Placebo — 25 mg po tid

SUMMARY:
The purpose of this study is to determine if sildenafil improves the exercise capacity and lung function of patients with chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Patients with chronic obstructive pulmonary disease (COPD) suffer from impaired exercise capacity and quality-of-life, largely related to shortness of breath. Many of the therapies currently available for COPD are aimed at improving these factors. Exercise capacity is limited in part by high blood pressure in the blood vessels in the lungs. Sildenafil, also known as Viagra, is an FDA-approved therapy for male erectile dysfunction. One of its effects is to relax (or open) the lung vessels, thereby lowering the blood pressure in the lungs. We hypothesize that sildenafil will result in an improvement in exercise capacity, quality-of-life, and shortness of breath.

Enrolled subjects will receive sildenafil or placebo for 4 weeks followed by exercise tests, breathing tests, and administration of quality-of-life questionnaires. Subjects will then receive placebo or sildenafil (whichever one they did not receive for the first 4 weeks) for another 4 weeks, followed by the same testing.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic obstructive pulmonary disease (COPD) or emphysema
* FEV1/FVC ratio < 70%
* FEV1 < 80%
* Stable medication regimen

Exclusion Criteria:

* COPD exacerbation or hospitalization in the past 3 months
* Heart disease
* Contraindication to sildenafil
* Unrelated lung disease
* Inability to walk or pedal on a stationary bike
* Pregnancy or breast-feeding
* Pulmonary hypertension at rest

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Kawut, M.D., M.S., Principal Investigator — Columbia University
Locations (1):
- Columbia Univeristy, College of Physicians and Surgeons, New York, New York, United States

REFERENCES:
- [Derived] Lederer DJ, Bartels MN, Schluger NW, Brogan F, Jellen P, Thomashow BM, Kawut SM. Sildenafil for chronic obstructive pulmonary disease: a randomized crossover trial. COPD. 2012 Jun;9(3):268-75. doi: 10.3109/15412555.2011.651180. Epub 2012 Feb 23. PMID 22360383

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period began in February 2005 and ended by November 2008.
Groups:
- Sildenafil /Placebo: 25 mg sildenafil is taken by mouth 3 times a day for 14 days followed by one week washout and then 25 mg placebo by mouth 3 times daily for 14 days.
- Placebo /Sildenafil: 25 mg placebo is taken by mouth 3 times a day for 14 days followed by one week washout and then 25 mg sildenafil by mouth 3 times daily for 14 days.
Period: Period 1: ( TREATMENT: 4 Weeks)
Arm/Group | Sildenafil /Placebo | Placebo /Sildenafil
Started | 6 | 4
Completed | 5 | 4
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Period 2 (WASHOUT: 1 Week)
Arm/Group | Sildenafil /Placebo | Placebo /Sildenafil
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0
Period: Period 3 ( TREATMENT: 4 Weeks)
Arm/Group | Sildenafil /Placebo | Placebo /Sildenafil
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Randomized Participants: All enrolled and randomized participants who were administered 25 mg Sildenafil and 25mg placebo at 2 different time periods.
Arm/Group | Randomized Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Secondary Outcome: Pulmonary Function FVC (Forced Vital Capacity)
Description: Data to calculate results for FVC was based on Period 1.
Time Frame: Period 1 (4 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: liters
Groups:
- Sildenafil: Sildenafil citrate 25 mg by mouth three times a day
- Placebo: Placebo by mouth three times a day.
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 6 | 4
liters | 2.8 [2.2 to 3.3] | 2.8 [2.2 to 3.3]

2. Primary Outcome: 6 Minute Walk Distance
Description: The distance a subject walked within 6 minutes was measured and documented.
Time Frame: Period 1 and Period 3 ( within 8 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: meters
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 10 | 9
meters | 458.2 [380 to 536] | 466.1 [388 to 544]

3. Primary Outcome: VO2 Peak (Oxygen Consumption at Peak Exercise)
Description: Oxygen consumption at peak exercise was measured at scheduled timepoints during treatment periods 1 and 3.
Time Frame: Period 1 and Period 3 ( within 8 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/kg/min
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 10 | 9
ml/kg/min | 13.7 [10.3 to 17.0] | 13.8 [10.3 to 17.3]

4. Secondary Outcome: Forced Expiratory Volume in the First Second (FEV1 )
Description: The volume of air exhaled in the first second. Data to calculate results for FEV1 was based on Period 1 only.
Time Frame: Period 1 ( 4 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: liters
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 6 | 4
liters | 1.1 [0.6 to 1.5] | 1.1 [0.7 to 1.6]

5. Secondary Outcome: Borg Dyspnea(Scale That Measures Breathlessness) Score at Finish of 6 Minute Walk Test (6MWT)
Description: Participants were asked to scale the breathlessness felt at the end of 6MWT from 0 to 10, with 0 being the least discomfort and 10 being the most discomfort in breathing.
Time Frame: Period 1 and Period 3 ( within 8 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Groups:
- Sildenafil: Group that received Sildenafil
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 10 | 9
Scores on a scale | 3.9 [2 to 5.9] | 3.8 [1.8 to 5.9]

6. Secondary Outcome: Diffusing Capacity of Carbon Monoxide (DLCO)
Description: Carbon Monoxide Diffusing Capacity was measured on the same days as the pulmonary function tests.
Time Frame: Period 1 and Period 3 ( within 8 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/min/torr
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 10 | 9
ml/min/torr | 11 [7.1 to 15] | 11 [7.1 to 15]

7. Secondary Outcome: Partial Pressure of Carbon Dioxide (PCO2) in Arterial Blood Gas (ABG)
Description: Partial pressure of carbon dioxide in ABG performed breathing room air at rest.
Time Frame: Period 1 and Period 3 ( within 8 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 10 | 9
mm Hg | 42 [38 to 45] | 40 [36 to 43]

8. Secondary Outcome: Partial Pressure of Oxygen (PO2) in Arterial Blood Gas (ABG)
Description: Partial Pressure of Oxygen in ABG breathing room air at rest.
Time Frame: Period 1 and Period 3 ( within 8 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 10 | 9
mm Hg | 73 [66 to 79] | 77 [71 to 84]

9. Secondary Outcome: A-a Gradient (Alveolar-arterial Gradient)
Description: A-a gradient was measured with ABG breathing room air at rest.
Time Frame: Period 1 and Period 3 ( within 8 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Groups:
- Placebo: Participants that received Placebo
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 10 | 9
mm Hg | 25 [19 to 33] | 23 [16 to 57]

10. Secondary Outcome: Oxygen Pulse
Description: Oxygen pulse during Cardiopulmonary exercise test at peak exercise.
Time Frame: Period 1 and Period 3 ( within 8 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/beat
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 10 | 9
ml/beat | 8.7 [6.4 to 11.0] | 9.5 [7.1 to 11.9]

11. Secondary Outcome: O2 Saturation at Peak Exercise
Description: O2 Saturation at Peak Exercise measured during the Cardiopulmonary exercise test.
Time Frame: Period 1 and Period 3 ( within 8 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of oxygen saturation
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 10 | 9
percentage of oxygen saturation | 95 [92 to 98] | 96 [93 to 99]

ADVERSE EVENTS:
Time Frame: 9 weeks
Description: Adverse events were monitored during the clinical trial period.
Groups:
- Sildenafil: 25 mg sildenafil is taken by mouth 3 times a day for 14 days followed by one week washout and then 25 mg placebo by mouth 3 times daily for 14 days.
- Placebo: 25 mg placebo is taken by mouth 3 times a day for 14 days followed by one week washout and then 25 mg sildenafil by mouth 3 times daily for 14 days.
Arm/Group | Sildenafil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 9/10 | 1/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil (N=10) | Placebo (N=9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Blurry vision (Eye disorders) | 3 | 0
Headache (General disorders) | 1 | 0
Pleuritic pain (General disorders) | 1 | 0
Nasal Congestion (General disorders) | 1 | 0
Upper respirartory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (General disorders) | 1 | 0
Rib Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Facial Flushing (General disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (General disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
The study had slow enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less